CLINICAL TRIAL: NCT04367961
Title: Auditory Profile and Language Development in Children Operated for Cleft Palate
Acronym: VELAUDI
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190493; 2019-A01660-57 (Other: ANSM)
Record Dates: First submitted 2020-04-26; First posted 2020-04-29 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-04

CONDITIONS: Deafness
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study about children with cleft palate from surgery to pre-adolescence :Description of language development and hearing profile.

DETAILED DESCRIPTION:
"Children with cleft palates are prone to complications that can impact on their overall development. Several factors such as serous otitis media or abnormal musculature of the velum can have consequences on hearing and language. In this context, it seems important to describe the evolution of this disease after surgery to better anticipate complications and improve their subsequent management. The aim of this study is to describe the hearing profile and language development of children with cleft palate from surgery to pre-adolescence. The hearing profile is assessed though an audiogram once or twice a year during the annual follow-up with the referring surgeon. Language development is assessed by the intelligibility scale, a validated questionnaire. This study will allow identification of : - predictive criteria for poor hearing and poor language development; - risk groups: type of cleft, medical history, genetic background, etc; - Level of speech disorder other than intelligibility: rhinolalia, eagerness for communication; - Other factors in the history of the disease: âge at surgery ; - history of chronic otitis media, ventilation tube placements; - nasalization and language disorder; - speech-language pathology; - History of hearing impairment; - age of first words; - Other ENT clinical history; - History of malformations; - Socio-economic level of the household; - Mother's language / number of languages spoken at home. This is a retrospective and prospective cohort study. Children aged 5 to 11 with a cleft palate operated on for a veloplasty at Robert Debré Hospital between 2008 and 2014 were included in the study between 2008 and 2014.

"

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5 to 11 years old operated on for a veloplasty at the Robert Debré Hospital
* operated between 2008 and 2014
* having a cleft veil with or without a cleft lip and palate

Exclusion Criteria:

* Children operated on for primary veloplasty outside the Robert Debré Hospital, and coming for secondary veloplasty.

Child operated on for a veloplasty for a cause other than the velar cleft.

Ages: 5 Years to 11 Years | Sex: All
Age Groups: Child
Study Population: Children with a cleft vein operated on for a veloplasty at Robert Debré Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-29 (Actual)

PRIMARY OUTCOMES:
The hearing profile is assessed though an audiogram once or twice a year during the annual follow-up with the referring surgeon. Language development is assessed by the intelligibility scale, a validated questionnaire | 1 day
  The hearing profile is assessed though an audiogram once or twice a year during the annual follow-up with the referring surgeon. The hearing test will be adapted depending the age of the child. Language development is assessed by the intelligibility scale, a validated questionnaire. The parent is answering the questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Debré Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided